CLINICAL TRIAL: NCT07256184
Title: Evaluation of Clinical, Pathologic, and Molecular Determinants of Prognosis and Treatment Response in Patients With Metastatic Malignant Melanoma: A Multicenter Retrospective Study
Brief Title: Prognostic and Treatment-Response Factors in Metastatic Melanoma: Multi-Center Analysis
Acronym: MEL-CARE
Status: Completed | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Galip Can Uyar, Medical Oncologist, Ankara Etlik City Hospital
Other Study IDs: AEŞH-BADEK-2025-0153; AEŞH-BADEK-2025-0153 (Other: Ankara Etlik City Hospital Scientific Research and Evaluation Ethics Committee)
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Malignant Melanoma
Keywords: melanoma; metastatic melanoma; prognosis; treatment response; immunotherapy; targeted therapy; BRAF mutation; PD-1 inhibitors; CTLA-4 inhibitors; dermatologic toxicity; adverse events
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multicenter Metastatic Melanoma Cohort: Includes adult patients diagnosed with metastatic malignant melanoma and treated between November 2022 and December 2024. Systemic therapies included immune checkpoint inhibitors (nivolumab, pembrolizumab, ipilimumab), BRAF/MEK targeted agents (dabrafenib, trametinib, vemurafenib, encorafenib, binimetinib), and chemotherapy (dacarbazine or temozolomide). Treatment was delivered per routine clinical practice; no experimental assignment occurred.
  Interventions: Drug: Systemic Therapy for Metastatic Melanoma

INTERVENTIONS:
Drug: Systemic Therapy for Metastatic Melanoma — Standard systemic treatments administered for metastatic malignant melanoma, including immune checkpoint inhibitors (nivolumab, pembrolizumab, ipilimumab), targeted therapy (dabrafenib, trametinib, vemurafenib, encorafenib, binimetinib), and chemotherapy (dacarbazine or temozolomide regimens). All treatments were provided as part of routine institutional clinical practice. No investigational or randomized assignment was performed. Treatment information was collected retrospectively from medical records for evaluation of prognostic and treatment-response outcomes.

SUMMARY:
This multicenter, retrospective observational study aims to identify clinical, pathological, and molecular factors associated with prognosis and treatment response in patients with metastatic malignant melanoma. Medical records of adult patients diagnosed and treated between November 2022 and December 2024 at participating oncology centers in Türkiye were reviewed.

Data collected include demographic features, disease characteristics, histopathologic findings, treatment modalities (immune checkpoint inhibitors, targeted therapy, or chemotherapy), and dermatologic adverse events. These variables will be analyzed in relation to survival outcomes to provide real-world evidence supporting personalized management strategies in metastatic melanoma.

DETAILED DESCRIPTION:
This multicenter retrospective cohort study evaluates clinical, pathological, and molecular factors that may influence prognosis and treatment response in patients with metastatic malignant melanoma treated between November 2022 and December 2024. The study focuses on routinely collected real-world data, including demographic characteristics, disease features, systemic treatment regimens, and dermatologic adverse events.

The primary analytical objectives are to assess associations between baseline variables and treatment outcomes, including Progression-Free Survival (PFS), Overall Survival (OS), and Objective Response Rate (ORR). Dermatologic and systemic toxicities graded using CTCAE v5.0 will also be explored for their potential impact on treatment continuity and outcomes. The study uses descriptive statistics, survival analyses, and Cox regression models. No experimental interventions are assigned, and all treatments were delivered as part of routine clinical practice.

This description provides an overview of study intent and analytic framework without duplicating detailed eligibility criteria or outcome definitions recorded in other submission fields.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically or cytologically confirmed metastatic malignant melanoma
* Received ≥1 line of systemic therapy
* Complete baseline and follow-up data
* At least one measurable lesion or clinical response assessment
* Managed between November 2022 - December 2024 at participating centers

Exclusion Criteria:

* Incomplete clinical or pathological data
* Uncertain or revised diagnosis
* Metastasis developing outside the inclusion window
* Another primary malignancy (except allowed types)
* Lost to follow-up before first response assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with metastatic malignant melanoma treated with standard systemic therapy, including immune checkpoint inhibitors, BRAF/MEK inhibitors, or chemotherapy. Data were extracted retrospectively from electronic medical records across multiple oncology centers in Türkiye.
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From treatment initiation to disease progression or death, up to December 2024.
  Progression-Free Survival (PFS) is defined as the time from initiation of systemic therapy to the earliest date of radiologically or clinically documented disease progression or death from any cause. Disease progression will be determined based on imaging studies or clinical evaluations recorded in medical files. Patients alive without documented progression at last follow-up will be censored.

SECONDARY OUTCOMES:
Overall Survival (OS) | From treatment initiation to death or last follow-up, up to December 2024.
  Overall Survival (OS) is defined as the time from systemic therapy initiation to death from any cause. Patients alive at last follow-up will be censored.
Objective Response Rate (ORR) | From treatment initiation to best documented response, within November 2022 - December 2024.
  Objective Response Rate (ORR) is defined as the proportion of patients achieving a Complete Response (CR) or Partial Response (PR) according to radiologic or clinical assessments documented in medical records. Responses will be determined by follow-up imaging or clinical examination.
Incidence of Dermatologic Adverse Events | From treatment initiation to last follow-up, up to December 2024.
  Incidence and grade of dermatologic adverse events, reported as number of patients (n) and percentage (%), including rash, pruritus, vitiligo, mucositis, and other toxicities graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Treatment Discontinuation Due to Toxicity | From treatment initiation to treatment discontinuation or last follow-up, up to December 2024.
  Proportion of patients who discontinued or interrupted systemic therapy due to treatment-related adverse events. Reasons and timing for discontinuation will be recorded based on medical records and categorized according to therapy type (immune checkpoint inhibitors, targeted therapy, or chemotherapy).
Disease Control Rate (DCR) | From treatment initiation to best documented response assessment, within November 2022 - December 2024.
  Disease Control Rate (DCR) is defined as the proportion of patients achieving Complete Response (CR), Partial Response (PR), or Stable Disease (SD) as their best overall documented response during systemic therapy. Determined through radiologic or clinical assessment.
Impact of Dermatologic Adverse Events on Progression-Free Survival | From treatment initiation to progression or last follow-up, up to December 2024.
  The association between dermatologic adverse events and PFS, expressed as a hazard ratio (HR) derived from survival analysis models.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara Etlik City Hospital, Ankara, Yenimahalle
  - Gazi University, Medical Oncology Department, Ankara, Çankaya

IPD SHARING:
Plan to Share IPD: No